CLINICAL TRIAL: NCT00889785
Title: Situational Problem Solving in Adolescents With Type 2 Diabetes: Enhancing an RCT
Brief Title: Situational Problem Solving in Adolescents With Type 2 Diabetes: Enhancing a Randomized Controlled Trial (RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Russell Rothman, Associate Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 090076; K23DK065294 (NIH); R03DK081726 (NIH)
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Adolescents With Type 2 Diabetes
Keywords: Adolescents; Type 2 Diabetes; Behavioral Research
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Usual Care) (Active Comparator): Patients will continue to review usual care in the diabetes clinic. Patients will receive monthly phone calls as an active control condition.
  Interventions: Behavioral: Usual Care
- Intervention (Experimental): The intervention will include participation in a comprehensive disease management program that includes: (1) application of treatment algorithms, (2) phone assessment from a diabetes nurse practitioner and dietician to assess barriers and promote problem solving, treatment adherence and management, and (3) a behavioral Internet-administered self-management problem solving component.
  Interventions: Behavioral: Comprehensive intervention (disease management program)

INTERVENTIONS:
Behavioral: Comprehensive intervention (disease management program) — The intervention will include participation in a comprehensive disease management program that includes: (1) application of treatment algorithms, (2) phone assessment from a diabetes nurse practitioner and dietician to assess barriers and promote problem solving, treatment adherence and management, and (3) a behavioral Internet-administered self-management problem solving component.
  Arms: Intervention
Behavioral: Usual Care — Will receive usual care and monthly phone calls as an active control.
  Arms: 1 (Usual Care)

SUMMARY:
The proposed research will test a new comprehensive disease management intervention with adolescents who have type 2 diabetes using a randomized controlled trial (RCT). Adolescents subjects with a history of Type 2 Diabetes and a parent caregiver will be consented, enrolled, and randomly assigned to either an 6-month intervention (N=44) or a "usual care" comparison (N=44). Recruitment will take place within the Vanderbilt Eskind Pediatric Diabetes Clinic. The intervention will include participation in a comprehensive disease management program that includes: (1) application of treatment algorithms, (2) phone assessment from a diabetes nurse practitioner and dietician to assess barriers and promote problem solving, treatment adherence and management, and (3) a behavioral Internet-administered self-management problem solving component. Outcomes include self-reported self-management behaviors (exercise, diet, medication adherence, etc.), blood pressure, weight/BMI, and glycated hemoglobin (A1C).

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of T2DM will be included if they are:

1. Age 12-19 years
2. A clinical diagnosis of T2DM (according to the patient and their health provider in the clinic)
3. Actively receive diabetes care in the Eskind Diabetes Clinic
4. Willingness of patient and a caregiver to access the Internet to complete problem solving activities
5. Adolescent address is the same as their primary caregiver participating in the study

Exclusion Criteria:

Patients will be excluded if they meet any of the following:

1. Identify an outside practitioner as the main provider of their diabetes care
2. Have a significant psychiatric illness such as severe depression or active psychosis that would impact on the ability to participate in the study
3. Life expectancy of <6 months
4. Unable to access the Internet from any convenient location
5. Blind or deaf

Parent Inclusion criteria:

1. Parents must be a primary caregiver of an adolescent with a diagnosis of T2DM between the ages 12-19 seen at the Eskind Clinic
2. Willingness of patient and a caregiver to access the Internet to complete problem solving activities.

Parent Exclusion criteria:

Patients will be excluded if they meet any of the following:

1. Identify an outside practitioner as the main provider of their child's diabetes care
2. Self report of significant psychiatric illness such as severe depression or active psychosis that would impact on the ability to participate in the study
3. life expectancy of <6 months
4. unable to access the Internet from any convenient location
5. blind or deaf.

Joint Inclusion criteria:

Both the primary caregiver (parent) and adolescent must agree to participate in the research.

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2009-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
A1C | 0,3,6 months
Lipids | 0,3,6 months

SECONDARY OUTCOMES:
blood pressure | 0,3,6 months
self-care behaviors | 0,3,6 months

CONTACTS AND LOCATIONS:
Overall Officials: Russell L Rothman, MD MPP, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Univ Medical Center, Nashville, Tennessee, United States